CLINICAL TRIAL: NCT06238674
Title: Early Goal Nutrition Therapy Guided by Indirect Calorimetry and Nitrogen Balance Among Critically Ill Patients With Acute Kidney Injury
Brief Title: Early Goal Nutrition Therapy Guided by Indirect Calorimetry and Nitrogen Balance Among Critically Ill Patients With Acute Kidney Injury (ENGINE Study)
Acronym: ENGINE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wankawee Jeerangsapasuk (Other)
Collaborators: Thammasat University Hospital (Other)
Responsible Party: Sponsor-Investigator, Wankawee Jeerangsapasuk, Clinical nephrology fellow, Principal Investigator, Doctor, Thammasat University
Organization: Thammasat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-IM-0-281/65
Record Dates: First submitted 2024-01-07; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Critically Ill; Nutrition Disorders; Acute Kidney Injury
Keywords: Indirect calorimetry, nutrition in acute kidney injury, nutrition in critically ill, nitrogen balance
MeSH Terms: conditions — Critical Illness; Nutrition Disorders; Acute Kidney Injury | interventions — Calorimetry, Indirect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualised energy and protein delivery guided by indirect calorimetry and nitrogen balance (Experimental): Energy delivery will be guided by indirect calorimetry with the aim to meet 70-100% of the most recent energy expenditure measurement and protein delivery guided by nitrogen balance with the aim to positive nitrogen balance with the maximum of 1.3 g/kg/d after 72 hours of admission and continue for total of 14 days by enteral or parenteral feeding routes
  Interventions: Other: indirect calorimetry and nitrogen balance
- Standard care nutrition (Active Comparator): Energy and protein delivery will be according to predictive equation estimates and usual site practice along enteral feeding
  Interventions: Other: Indirect calorimetry (Standard care nutrition arm)

INTERVENTIONS:
Other: indirect calorimetry and nitrogen balance — nutrition therapy with energy guided by indirect calorimetry measurements and total protein guided by nitrogen balance with the maximum of 1.3 g/kg/d
  , repeated indirect calorimetry if renal replacement therapy was initiated and follow up of urea nitrogen balance after 7 days of intervention to guarantee positive nitrogen balance
  Other Names: Metabolic demand
  Arms: Individualised energy and protein delivery guided by indirect calorimetry and nitrogen balance
Other: Indirect calorimetry (Standard care nutrition arm) — indirect calorimetry measurements using the Q-NRG+ device will be conducted and urea nitrogen balance were measured . In the standard care nutrition arm, clinicians will be blinded to indirect calorimetry and urea nitrogen balance measurements
  Arms: Standard care nutrition

SUMMARY:
The goal of this clinical trial is to investigate the effects of nutrition therapy guided by indirect calorimetry and nitrogen balance among critically ill patients with acute kidney injury. The main question it aims to answer whether nutrition therapy guided by indirect calorimetry and nitrogen balance could improve 28 days mortality among critically ill patients with acute kidney injury or not.

type of study: clinical trial Participants will be provided enteral or parenteral nutrition after randomization(48-72 days after admissions) with total energy guided by indirect calorimetry measurements and total protein by nitrogen balance with maximum of 1.3 gram per kilogram per day for total of 14 days If there is a comparison group: Researchers will compare with the control groups (nutrition therapy provided by physician using clinical equation of choice or judgements to see if participants were provided with these interventions, their 28 days mortalities would be better

DETAILED DESCRIPTION:
The gold standard for determining energy requirements was recommended by the European Society for Parenteral and Enteral Nutrition (ESPEN) guideline 2021 to use indirect calorimetry(IC), a noninvasive method that allows resting energy expenditure (REE) evaluation based on measurements of oxygen consumption and carbon dioxide production in the exhaled air.

As there are no high-quality studies that investigated energy and protein provision in hospitalized patients with acute kidney injury(AKI) or Acute kidney disease (AKD), the recommendations were based on the guidelines and clinical trials from critically ill and polymorbid internal medicine patients because these guidelines and trials included patients with kidney disease.

Moreover, there were clinical trials in critically ill patients with severe acute kidney injury found the varying of metabolic states among these patients categorized by IC measurements and no association between calorie intake and mortality outcome.

Even though the aforementioned researches did not suggest a link between calorie intake and mortality outcome, no studies were able to meet the energy targets set using indirect calorimetry measurements.

This study aims to prove the necessary and benefit of early nutrition therapy after 72 hours of admission with total energy guided by indirect calorimetry measurements aims to meet 70-100% from measurements and total protein guided by urine urea nitrogen balance aims to positive nitrogen balance with maximum of 1.3 gram per kilogram of actual body weight per day for total of 14 days on survival & renal outcomes in critically ill patients with acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years old
* Mechanically ventilated patients with acute kidney injury by Kidney Disease Improving Global Outcomes (KDIGO) criteria
* Expected length of ICU stay more than 72 hours and accept to follow the study protocol

Exclusion Criteria:

* Underlying chronic kidney disease stage 4 or 5 according to KDIGO staging
* received renal replacement therapy prior to admission
* Post cardiothoracic surgery
* Required fraction of inspired oxygen inspired oxygen fraction (FiO2) more than 0.6
* Pregnancy
* BMI below 17 or above 35 kg/m2 or very high risk refeeding syndrome
* Cirrhosis Child-Pugh score C

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-28 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | up to 28 days after randomization
  28 day mortality

SECONDARY OUTCOMES:
length of ICU stay | up to 28 days
  Duration of ICU stay (days)
ICU mortality | up to 28 days
  ICU mortality
Rate of new renal replacement therapy | up to 28 days
  Rate of new renal replacement therapy (times)
Peak serum creatinine | up to 28 days
  Peak serum creatinine (mg/dl)
Nosocomial infection | up to 28 days
  incident of Nosocomial infection (yes or No)
Blood sugar level and amount of insulin usage | up to 28 days
  average amount of daily amount of insulin usage (unit)
60 day mortality | up to 60 days
  60 day mortality
Duration of mechanical ventilation | up to 28 days
  Duration of mechanical ventilation (days)
Treatment separation in energy adequacy | up to 28 days
  Energy adequacy % will be calculated as energy delivery (kcal)/ measured energy expenditure (kcal) and expressed as a percentage
adverse events | up to 28 days
  feeding intolerance, diarrhea (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Wankawee Jeerangsapasuk, Bachelor, Study Director — Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Rangsit City Municipality, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data sharing requests will be considered following publication of the primary trial data on an individual basis by the trial management committee (the data custodians). Data sharing will only be considered for investigator-initiated, independent researchers who provide a written data evaluation proposal that is judged to be methodologically sound. A data sharing agreement will be required to detail conditions under which data is shared and used. Resulting publications should appropriately cite and acknowledge the original data custodians. Requests for data sharing are to be made to wankaweej@gmail.com and the corresponding author, Dr Aphichat Chatkrailert; tengaphi@gmail.com
Supporting Information: Study Protocol, CSR
Access Criteria: depend on responsible party agreements

REFERENCES:
- [Background] Susantitaphong P, Cruz DN, Cerda J, Abulfaraj M, Alqahtani F, Koulouridis I, Jaber BL; Acute Kidney Injury Advisory Group of the American Society of Nephrology. World incidence of AKI: a meta-analysis. Clin J Am Soc Nephrol. 2013 Sep;8(9):1482-93. doi: 10.2215/CJN.00710113. Epub 2013 Jun 6. PMID 23744003
- [Background] Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten H, Ronco C, Kellum JA. Continuous renal replacement therapy: a worldwide practice survey. The beginning and ending supportive therapy for the kidney (B.E.S.T. kidney) investigators. Intensive Care Med. 2007 Sep;33(9):1563-70. doi: 10.1007/s00134-007-0754-4. Epub 2007 Jun 27. PMID 17594074
- [Background] Fiaccadori E, Sabatino A, Barazzoni R, Carrero JJ, Cupisti A, De Waele E, Jonckheer J, Singer P, Cuerda C. ESPEN guideline on clinical nutrition in hospitalized patients with acute or chronic kidney disease. Clin Nutr. 2021 Apr;40(4):1644-1668. doi: 10.1016/j.clnu.2021.01.028. Epub 2021 Feb 9. PMID 33640205